CLINICAL TRIAL: NCT00849394
Title: An Evaluation of Proteinuria in Patients Receiving Shortened Infusions of Bevacizumab
Brief Title: Evaluation of Protein in the Urine in Patients Receiving Bevacizumab
Status: Completed | Type: Observational
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sachin Shah, Pharm.D., BCOP, Texas Tech University Health Sciences Center School of Pharmacy
Other Study IDs: 07-097; 122007-001;; A07-3423
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2009-02

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: bevacizumab; proteinuria
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Shortened infusions of bevacizumab

SUMMARY:
This is a clinical research study to look at the incidence of proteinuria (a condition in which urine contains an abnormal amount of protein) caused by shortened infusions (given into the vein over 10 or 15 minutes) of bevacizumab (a medication prescribed for colon, lung, or breast cancer). There are currently no published studies or clinical data looking at how safe shortened infusions of bevacizumab are in relationship to the side effect of proteinuria. We hypothesis that shortened infusions of bevacizumab will result in an increased risk for proteinuria compared to the standard infusions of this agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years older
* Patients must be receiving his/her first dose of bevacizumab
* Patients must sign an informed consent

Exclusion Criteria:

* Patients receiving > 10 mg/kg doses of bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 106 patients receiving bevacizumab doses of < 10 mg/kg at a rate of 0.5 mg/kg/min in hematology/oncology outpatient clinic. Most of the patients are likely to have advanced stage colon or rectal cancer.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2007-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of shortened infusions (0.5 mg/kg/min) of bevacizumab on the incidence of proteinuria. | 3-6 months

SECONDARY OUTCOMES:
To evaluate the time (number of days) to the incidence of proteinuria with shortened infusions of bevacizumab AND to evaluate the effect of controlled versus uncontrolled hypertension and the incidence of proteinuria. | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Shah, Pharm.D., Principal Investigator — Texas Tech University Health Sciences Center School of Pharmacy
Locations (3):
- United States (3):
  - VA North Texas Health Care System, Dallas, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas